CLINICAL TRIAL: NCT01298791
Title: The Impact Of Physician Communication On Family Inpatient Experience
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit participants
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Michael Silverstein, BMC Attending Physician, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 34423
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Parental/Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction | interventions — Sitting Position; Standing Position

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Provider sitting (Experimental): Providers seated during communication through hospitalization
  Interventions: Behavioral: Sitting
- Provider standing (control) (Experimental): Providers standing during communication through hospitalization
  Interventions: Behavioral: Standing

INTERVENTIONS:
Behavioral: Sitting — Providers will sit during inpatient family-centered walk rounds throughout the communication during rounds. The participating members of the care team (attending physician, resident and medical student) will remain seated while communicating with the patient and caregiver.
  Arms: Provider sitting
Behavioral: Standing — Providers will stand during inpatient family-centered walk rounds throughout the communication during rounds. The participating members of the care team (attending physician, resident and medical student) will remain standing while communicating with the patient and caregiver.
  Arms: Provider standing (control)

SUMMARY:
Patient satisfaction is affected by physician communication styles and communication at the bedside. The investigators are conducting a randomized controlled trial involving both providers and families to determine if providers sitting down while talking with families, will improve one aspect of quality care delivered during an inpatient stay as measured by patient/family satisfaction. The investigators will additionally study the affects of the intervention on the following outcomes: family assessment of provider communication, readmission rates, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Providers: all attendings, residents, and medical students involved in the care of patients on the pediatric inpatient wards during the study period.
* Families (Parents or legal guardians and children):
* (1) inpatient admissions to the pediatrics medical service at Boston Medical Center
* (2) whose parents or guardian have agreed to participate in family centered walk rounds
* (3) patients age 17 or younger who have family members present at the bedside each morning of hospitalization
* (4) English speaking.

Exclusion Criteria:

* (1) All patients/families that as part of admission justification involves social assessment and concern by the patient care team, including patients with neonatal abstinence syndrome, child maltreatment, and concern for neglect.
* (2) All patients transferred to or from PICU as part of their inpatient care
* (3) All patients transferred from an outside institution to the inpatient ward for further care secondary to progression of disease.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Estimated); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Patient/family satisfaction | 4mo
  Questionnaire obtains basic provider information
Patient/family Satisfaction | 4 mo
  Caregiver questionnaire obtains baseline information on caregiver and patients
Patient/family satisfaction | 4 months
  PSQ-18: Assesses parental satisfaction with medical care

SECONDARY OUTCOMES:
Length of stay | 4 months
  Chart review of length of inpatient hospitalization during intervention
Readmission rate | 5 mo
  Chart review and parental contact regarding readmission for same reason of initial hospitalization
Family discharge preparedness | 4 mo
  Brief PREPARED instrument
Follow-up appointment attendance | 5 mo
  Chart review and communication with caregivers regarding keeping follow-up appointment
Family assessment of doctor-patient communication skills | 4 mo
  Crossley Communication Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverstein, MD, MPH, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States